CLINICAL TRIAL: NCT04402567
Title: "Showing the Truth": Impact and Burden of Rugby Injuries in Argentina. A Complete Season Retrospective Multicentric Study.
Brief Title: Impact and Burden of Rugby Injuries in Argentina. A Complete Season Retrospective Multicentric Study.
Acronym: ARugby
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Donación Francisco Santojanni (Other)
Responsible Party: Principal Investigator, Mauro Andreu, Prof. Lic. Klgo. Ftra. Mauro Andreu, Hospital Donación Francisco Santojanni
Other Study IDs: HGADFS19052020-01
Record Dates: First submitted 2020-05-17; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Injuries
Keywords: epidemiology; Incidence; Injury severity; Football
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — Not Apply

SUMMARY:
The aim of this study was to describe the prevalence, incidence and injury load suffered in male amateur rugby players from Argentina during a competitive season in 2019.

DETAILED DESCRIPTION:
Introduction:

Currently, Rugby is a sport that is giving priority to the well-being of the player. Players are subjected to high training and match loads exposing them to constant stress that can lead to overload injuries in addition to frequent contact injuries. Despite knowing what the situation is like at the international and national level, the "Unión Argentina de Rugby" lacks conclusive epidemiological data.

Our main purpose was to describe the prevalence, incidence and injury load suffered in male amateur rugby players from Argentina during a competitive season in 2019.

Design:

Observational, descriptive, retrospective and multicenter study.

Participants:

250 male amateur rugby players belonging to three clubs from three rugby unions (Buenos Aires, Córdoba and Rosario) of Argentina.

Methods:

Registration methods were applied according to the consensus of the World Rugby by a single observer per center. Injuries occurred in players from top rosters of 3 amateur rugby clubs (data collection centers) as well as the number of matches and hours of training were recorded. Medical diagnoses were classified under the rules of the OSIICS classification system. The incidence (injuries / 1000 hours-game-player), prevalences (point and period), the severity (days of absence) and the injury load will be calculated as well as the location, type, nature. This study followed the guidelines of the STROBE-SIIS Initiative Declaration.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Participation in more than 80% during training and matches of the competitive season.
* First, intermediate, Pre-intermediate A and Pre-intermediate B categories of the University teams of Córdoba, Old Resian and Los Matreros, belonging to UAR member unions.

Exclusion Criteria:

- Lost patient data

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male Argentine amateur rugby players of the 2019 season
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-05-20 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Injury Incidence | 9 months
  injuries/1000 hours-player

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Andreu, BSc, Study Director — Hospital Donación Francisco Santojanni

IPD SHARING:
Plan to Share IPD: Undecided